CLINICAL TRIAL: NCT03934255
Title: Central and Peripheral Circadian Mechanisms Underlying Non-Dipping Blood Pressure in Blacks
Brief Title: Circadian Mechanisms Underlying Non-Dipping Blood Pressure in Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Stephen Justin Thomas, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300003266
Record Dates: First submitted 2019-04-19; First posted 2019-05-01 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Circadian Rhythm; Blood Pressure

STUDY DESIGN:
Intervention Model Description: Constant routine protocol in Blacks with dipping and non-dipping blood pressure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Constant Routine Protocol (Experimental): Participants will be kept in constant conditions for 30 hours to observe circadian physiology in the absence of light, physical activity, and meals.
  Interventions: Other: Constant Routine Protocol

INTERVENTIONS:
Other: Constant Routine Protocol — Constant routine protocols are used in circadian research to examine underlying circadian rhythms in the absence of light, activity, and meals

SUMMARY:
This study seeks to examine central and peripheral circadian mechanisms in Blacks with appropriately dipping systolic blood pressure (blood pressure that dips by at least 10%) compared with non-dipping systolic blood pressure (blood pressure that dips by less than 10%) using a constant routine protocol. Constant routine protocols are commonly used in the field of circadian biology to examine rhythms in biological processes while controlling the entraining effects of light, activity, and diet.

DETAILED DESCRIPTION:
This study will enroll a total of 40 participants (n=20 non-dippers; n=20 dippers) to complete a 30-hour constant routine protocol. Participants will undergo baseline testing that includes anthropometric measurements, clinic blood pressure measurements, completion of self-report questionnaires on sleep and mood, be fitted with an ambulatory blood pressure monitor and actigraphy watch, and be provided with home sleep testing (HST) equipment.

Following completion of baseline assessment, eligible participants will be scheduled for the 30-hour constant routine protocol. The 30-hour constant routine protocol will allow for the hourly collection of saliva, collection of buccal cells every 4 hours, and constant monitoring of core body temperature, all of which are primary outcomes in the assessment of central and peripheral circadian clock markers. Amplitude and phase of these outcomes will be assessed in non-dippers versus dippers.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American race
* Age 18 years or older

Exclusion Criteria:

* Work alternating or night shifts
* Pregnant or nursing
* Current illicit drug use
* History of severe mental illness
* Medical conditions that would be contraindicated for a constant routine protocol
* Take anti-hypertensive medications or beta-blockers
* Severe obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Melatonin phase | Melatonin phase during a 30-hour constant routine protocol
  Circadian phase of melatonin obtained from saliva
Melatonin amplitude | Melatonin amplitude during a 30-hour constant routine protocol
  Circadian amplitude of melatonin obtained from saliva
Core body temperature phase | Core body temperature phase during a 30-hour constant routine protocol
  Circadian phase of core body temperature recorded and transmitted wirelessly
Core body temperature amplitude | Core body temperature amplitude during a 30-hour constant routine protocol
  Circadian amplitude of core body temperature recorded and transmitted wirelessly
Buccal cell mRNA expression | Expression of Bmal1 and Period 3 during a 30-hour constant routine protocol
  Expression of Bmal1 and Period 3 obtained from buccal cell mRNA

SECONDARY OUTCOMES:
Cortisol phase | Cortisol phase during a 30-hour constant routine protocol
  Circadian phase of cortisol obtained rom saliva
Cortisol amplitude | Cortisol amplitude during a 30-hour constant routine protocol
  Circadian amplitude of cortisol obtained rom saliva

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Details regarding sharing IPD are undecided. Protocols and consent forms will be shared. Requests may be made to the study PI.